CLINICAL TRIAL: NCT00848835
Title: Long Term Integrity Follow-up Evaluation
Acronym: LEAD LIFE
Status: Completed | Type: Observational
Sponsor: Guidant Corporation (Industry)
Responsible Party: Anne Swearingen, Boston Scientific
Other Study IDs: LEAD LIFE
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Sudden Cardiac Death
Keywords: defibrillator
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- control: all patients in the control group
  Interventions: Device: defibrillation lead (ENDOTAK EZ and RELIANCE)

INTERVENTIONS:
Device: defibrillation lead (ENDOTAK EZ and RELIANCE) — defibrillation lead

SUMMARY:
To document the performance of the Guidant ENDOTAK EZ and the RELIANCE defibrillation leads over 5 years.

DETAILED DESCRIPTION:
There are few prospective long term follow-up studies on implanted cardiac device (pacemaker/implantable cardioverter defibrillator (ICD)) survivability. This study will evaluate the long term performance (5 years) of the transvenous defibrillation leads (ENDOTAK ENDURANCE EZ and teh ENDOTAK RELIANCE. Data will be collected at implant, 1 and 6 months, 1,3 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients selected for Guidant ICD system implant, available for follow-up at the defined intervals

Exclusion Criteria:

* Patients enrolled in other studies, not available for follow-up, < 18 yrs, unable to sign consent, life expectancy < 1 year due to a medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients who are indicated for a market released ICD
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2002-03; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Sterns, MD, Principal Investigator — Victoria Cardiac Arrythmia trials